CLINICAL TRIAL: NCT06172426
Title: Incidence of Psoriatic Arthritis Among Psoriasis Patients Newly Initiated With Secukinumab in a US Claims Database and a UK Registry
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAIN457A2026
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Psoriatic Arthritis; Psoriasis
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- MarketScan® secukinumab, other biologics/apremilast, and any biologics/apremilast cohort
- BADBIR secukinumab cohort

SUMMARY:
This was a retrospective cohort study to assess the incidence rate of psoriatic arthritis (PsA) among psoriasis (PsO) patients newly initiated on secukinumab or any biologics/apremilast (small molecule). The analysis was performed in two databases, IBM® MarketScan® database: Commercial Claims and Encounters (CCAE) and Medicare Supplemental Beneficiaries (MDCR) from 01 January 2010 to 30 June 2021 and BADBIR from 01 January 2016 to 01 September 2021.

ELIGIBILITY:
MarketScan® secukinumab cohort:

Inclusion criteria:

* Included patients with at least 1 secukinumab claim between 01 January 2015 and 30 June 2020 (index date is the first secukinumab claim)
* Included patients age ≥18 years as of the year of index date
* Included patients with at least 1 non-ruleout psoriasis diagnosis during 2 years of pre-index period
* Included patients with continuous medical/pharmacy coverage in the 2-year pre-index period
* Included patients with continuous medical/pharmacy coverage in the 1-year post-index period

Exclusion criteria:

* Excluded patients with any psoriatic arthritis diagnosis during 2 years to 5 years pre-index period, as well as on the index date
* Excluded patients with any biologics/apremilast including secukinumab claim during the 2-year pre-index (excluding index date)
* Excluded patients received other non-secukinumab biologics/apremilast during 6 months post index date period (including index date) (This criterion is only applicable for the secukinumab cohort)

BADBIR cohort:

Inclusion criteria:

* Included non-switched patients with secukinumab treatment on or after the enrollment between 01 January 2017 to 01 September 2020

  * Non-switched patients are those who did not use other biologics/apremilast treatments on the enrollment date
  * Index date will be the date of the first secukinumab treatment date
* Included patients with age ≥ 18 on the index date
* Included patients with psoriasis diagnosis in the pre-index period and index date
* Included patients with ≥ 1 year follow-up period

  * Follow-up period is the gap between patient's last visit date and index date

Exclusion criteria:

* Excluded patients with psoriatic arthritis (PsA) prior to and on index date
* Excluded patients with any biologics/apremilast including secukinumab in the baseline period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 1171 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Exposure-adjusted incidence rate of PsA per 100 patient-years among PsO patients who newly initiated secukinumab | Up to 11.5 years

SECONDARY OUTCOMES:
Time from secukinumab initiation to the first PsA diagnosis | Up to 11.5 years
Age | Baseline
Gender | Baseline
Region | Baseline
Insurance type | Baseline
Ethnicity | Baseline
Weight | Baseline
Height | Baseline
Body mass index (BMI) | Baseline
Prior treatments | Baseline
Hard-to-treat locations | Baseline
Comorbidities | Baseline
Dermatology Life Quality Index (DLQI) | Baseline
  The DLQI is a validated, 10-question, self-reported questionnaire to evaluate the patient's perception of the impact of skin disease on quality of life. The DLQI is rated on a 4-point scale (0 = not at all to 3 = very much). The highest possible total score for the DLQI is 30, and higher scores indicate more severe impact on quality of life.
Health Assessment Questionnaires - Disability Index (HAQ-DI) | Baseline
  The HAQ-DI is a 20-question scale assessing functional ability. The final HAQ-DI score ranges from 0 (no problems functioning) to 3 (not able to function).
Psoriasis Area and Severity Index (PASI) | Baseline
  The Psoriasis Area and Severity Index (PASI) is the most widely used tool for the measurement of severity of psoriasis. PASI combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease).
Body Surface Area (BSA) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, Basel, Switzerland